CLINICAL TRIAL: NCT05323175
Title: Can Erector Spinae Plane (ESP) Block Better Relieve Acute Renal Colic Pain Than Standard of Care
Brief Title: Erector Spinae Plane (ESP) Block for Renal Colic
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Michael Secko, MD, Clinical Associate Professor, Emergency Department, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB2021-00518
Record Dates: First submitted 2021-10-08; First posted 2022-04-12 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Renal Colic
Keywords: Erector spinae plane block
MeSH Terms: conditions — Renal Colic | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: Standard of care group + sham normal saline ESP block vs Standard of care + Ropivacaine ESP nerve Block group
Who Masked: Participant
Masking Description: Participant will not know which type of block they receive
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ESP Nerve Block for Renal colic (Active Comparator): On top of receiving standard of care, At T8 nerve level, with ultrasound guidance to bathe the nerve
  Interventions: Drug: Ropivacaine injection
- Standard of care (Active Comparator): Whatever medications the clinician normally treats renal colic with
  Interventions: Other: Standard of care medications

INTERVENTIONS:
Drug: Ropivacaine injection — Local anesthesia injected under ultrasound guidance
  Arms: ESP Nerve Block for Renal colic
Other: Standard of care medications — Whatever the ED clinicians normally give for renal colic pain
  Arms: Standard of care

SUMMARY:
Comparing standard of care to erector spinae plane block for acute renal colic pain.

DETAILED DESCRIPTION:
Will compare at times 0, 10 minute, 20 minute, 40 minute and 60 minutes after local nerve block given.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years old
* ASA Level I and II
* flank pain concerning for renal colic in ED

Exclusion Criteria:

* pregnant women
* subjects unable to appreciate ESP block landmarks under ultrasound
* skin infection over needle site insertion
* Allergy to local anesthesia (lidocaine/Ropivacaine)
* bleeding disorders
* serious cardiac, lung, liver or kidney dysfunction
* history of spine surgery
* history of spinal infection
* history of epidural injection within 6 months
* acute exacerbation of serious mental disease
* unable to consent
* unable to communicate pain level

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Baseline Pain before intervention | Before the ESP Block
  Using the Visual Analog Scale for Pain Assessment Tool with 0 meaning "No pain" and 10 meaning "Unbearable Pain"
Pain score at 10 minutes | 10 minutes after the ESP Block
  Using the Visual Analog Scale for Pain Assessment Tool with 0 meaning "No pain" and 10 meaning "Unbearable Pain"
Pain score at 20 minutes | 20 minutes after ESP Block
  Using the Visual Analog Scale for Pain Assessment Tool with 0 meaning "No pain" and 10 meaning "Unbearable Pain"
Pain score at 40 minutes | 40 minutes after ESP Block
  Using the Visual Analog Scale for Pain Assessment Tool with 0 meaning "No pain" and 10 meaning "Unbearable Pain
Pain score at 60 minutes | 60 minutes after ESP Block
  Using the Visual Analog Scale for Pain Assessment Tool with 0 meaning "No pain" and 10 meaning "Unbearable Pain

SECONDARY OUTCOMES:
Need for extra opiates | Starting from time 0 after the ESP Block intervention completed till discharge or urology intervention
  Record how much opioids patients receives starting after the ESP Block for both the "standard of care" patients and the ESP Block group

CONTACTS AND LOCATIONS:
Overall Officials: Michael Secko, MD, Principal Investigator — StonyBrook University Hospital
Locations (1):
- StonyBrook University Hospital, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aydin ME, Tekin E, Ahiskalioglu EO, Ates I, Karagoz S, Aydin OF, Ozkaya F, Ahiskalioglu A. Erector spinae plane block vs non-steroidal anti-inflammatory drugs for severe renal colic pain: A pilot clinical feasibility study. Int J Clin Pract. 2021 Mar;75(3):e13789. doi: 10.1111/ijcp.13789. Epub 2020 Nov 9. PMID 33099855